CLINICAL TRIAL: NCT01184599
Title: A Prospective Study of the Kidney Protective Effect of Aliskiren in Hypertensive Patients With IgA Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kagawa University (Other)
Responsible Party: Hirofumi Hitomi, Kagawa University, Faculty of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCGH-746
Record Dates: First submitted 2010-08-16; First posted 2010-08-19 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-05

CONDITIONS: Glomerulonephritis, IGA; Hypertension
Keywords: Aliskiren; Albuminuria; Angiotensinogen; collagen type IV; Transforming Growth Factor beta; aldosterone; renin; prorenin receptor; des-angiotensin I renin substrate; oxidative stress; advanced glycosylation end-product receptor; N,N-dimethylarginine
MeSH Terms: conditions — Glomerulonephritis, IGA; Hypertension; Albuminuria; Camurati-Engelmann Syndrome | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aliskiren — 150 mg/day p.o.

SUMMARY:
The purpose of this study is to evaluate the effect of aliskiren, a novel direct rennin inhibitor, on renal function and progress of renal disease in hypertensive patients with IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* IgA nephropathy confirmed by renal biopsy
* Hypertension (<= 125/75 mmHg)

Exclusion Criteria:

* Patients who have been treated with angiotensin type 1 receptor blocker or angiotensin-converting enzyme inhibitor within 4 weeks
* Severe hypertension (<= 180/110 mmHg) or secondary hypertension
* Patients with history of allergy or adverse effect for aliskiren
* Renal dysfunction (estimated Glomerular Filtration Rate < 60 mL/min/1.73m2)
* Pregnancy
* Patient treated with cyclosporine
* Hyperkalemia (serum potassium >= 5.6 mmol/L)
* Autoimmune disease including systemic lupus erythematosus
* Patients inadequate for the study

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Renal function (Creatinine clearance) | One year (every 6 months)
Urinary protein | One year (every 6 months)

SECONDARY OUTCOMES:
Urinary angiotensinogen | One year (every 6 months)
Urinary type 4 collagen | One year (every 6 months)
Urinary Transforming growth factor-beta | One year (every 6 months)
High-sensitivity C-reactive protein | One year (every 6 months)
Plasma Rennin Activity | One year (every 12 months)
Aldosterone | One year (every 12 months)
Asymmetric dimethylarginine | One year (every 12 months)
Advanced glycation end product | One year (every 12 months)
(Pro)renin receptor | One year (every 12 months)
Oxidative stress | One year (every 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Masahito Imanishi, Principal Investigator — Osaka City General Hospital
Locations (4):
- Japan (4):
  - Kurume University, School of Medicine, Fukuoka
  - Department of Internal Medicine, Osaka City General Hospital, Osaka
  - Ohno memorial Hospital, Osaka
  - Kinki University, Faculty of Medicine, Osaka